CLINICAL TRIAL: NCT00295932
Title: A Phase II Study of the Novel Proteasome Inhibitor Bortezomib in Combination With Rituximab, Cyclophosphamide and Prednisone in Patients With Relapsed/Refractory Indolent B-Cell Lymphoproliferative Disorders and Mantle Cell Lymphoma (MCL)
Brief Title: Bortezomib, Rituximab, Cyclophosphamide, and Prednisone in Treating Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other); Columbia University (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-103; MSKCC-05103; NCT00859443 (obsolete NCT alias)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-03

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; Waldenstrom macroglobulinemia; recurrent mantle cell lymphoma; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; Cyclophosphamide; Prednisone

ARMS (2):
- Arm I (Experimental): Patients receive cyclophosphamide IV and rituximab IV on day 1, oral prednisone on days 2-6, and bortezomib IV (at the MTD determined in phase I) on days 2, 5, 9, and 12. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: cyclophosphamide; Drug: prednisone
- Arm II (Experimental): Patients receive cyclophosphamide IV and rituximab IV on day 1, oral prednisone on days 2-6, and bortezomib IV (at the MTD determined in phase I) on days 2 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: cyclophosphamide; Drug: prednisone

INTERVENTIONS:
Biological: rituximab — Given IV
Drug: bortezomib — Given IV
Drug: cyclophosphamide — Given IV
Drug: prednisone — Given orally

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with cyclophosphamide, prednisone, and rituximab may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of bortezomib when given together with cyclophosphamide, prednisone, and rituximab and to see how well it works in treating patients with relapsed or refractory indolent B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bortezomib when given in combination with rituximab, cyclophosphamide, and prednisone (R-CP) in patients with relapsed or refractory indolent B-cell lymphoproliferative disorders or mantle cell lymphoma. (phase I)
* Determine the frequency and duration of complete and partial responses in patients treated with two different treatment regimes. (phase II)

Secondary

* Evaluate the progression-free survival, event-free survival, and overall survival of patients treated with this regimen. (phase II)
* Evaluate the toxicity profile of this regimen.

OUTLINE: This is a phase I dose-escalation study of bortezomib followed by a phase II randomized, multicenter study. Patients in phase II are stratified according to disease (mantle cell lymphoma vs indolent B-cell lymphoproliferative disorder vs transformed lymphoma).

* Phase I: Patients receive cyclophosphamide IV and rituximab IV on day 1, oral prednisone on days 2-6, and bortezomib IV on days 2 and 7. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive cyclophosphamide IV and rituximab IV on day 1, oral prednisone on days 2-6, and bortezomib IV (at the MTD determined in phase I) on days 2, 5, 9, and 12. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive cyclophosphamide IV and rituximab IV on day 1, oral prednisone on days 2-6, and bortezomib IV (at the MTD determined in phase I) on days 2 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month, every 4 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Chronic lymphocytic leukemia (CLL)
  * B-cell small lymphocytic leukemia (SLL)
  * Any marginal zone lymphoma
  * Grade 1-3A follicular lymphoma
  * Waldenstrom's macroglobulinemia
  * Mantle cell lymphoma
* No transformed indolent lymphoma
* Assessable disease (phase I)
* Measurable disease (phase I and II), defined as ≥ one lesion that can be accurately measured in ≥ 1 dimension as ≥ 2 cm by conventional techniques OR ≥ 1 cm by spiral CT scan

  * Lymph nodes measuring ≤ 1 cm in the short axis are considered normal
* Relapsed or refractory disease

  * Must have received at least 1 prior therapeutic regimen but no more than 3 prior conventional cytotoxic therapy regimens
* No known brain metastases or meningeal disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status > 50%
* Absolute neutrophil count > 1,000/mcl (more than 500/mcl if known lymphomatous involvement)
* Platelet count ≥ 50,000/mcl
* Total bilirubin < 1.5 times upper limit of normal (ULN) (less than 5 mg/dL if known history of Gilbert's disease)
* AST and ALT ≤ 2.5 times ULN (4 times ULN if liver involvement)
* Creatinine < 1.5 times ULN OR creatinine clearance > 50 mL/min
* Patients may have febrile episodes up to 38.5ºC without evidence of active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No New York Heart Association class III or IV congestive heart failure
* No uncontrolled intercurrent illness, including any of the following:

  * Ongoing or active infection
  * Cerebrovascular accident or transient ischemic attack within 6 months of study entry
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * EKG evidence of acute ischemia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No uncontrolled hypertension requiring active manipulation of antihypertensive medications
* No known or active HIV infection
* No history of hypersensitivity to bortezomib, boron, or mannitol
* No peripheral neuropathy > grade 2
* No other malignancy within the past 5 years except curatively treated non life-threatening malignancies, such as cutaneous basal cell or squamous cell carcinoma or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* Prior stem cell transplantation allowed

  * Preparative cytoreductive and high-dose therapies considered 1 prior therapy
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks since prior nitrosoureas or mitomycin C)
* At least 12 weeks since prior radioimmunotherapy

  * One prior course comprising tositumomab or ibritumomab tiuxetan allowed
* At least 1 week since prior palliative steroids for NHL
* No therapeutic monoclonal antibodies (e.g., rituximab, tositumomab, ibritumomab, alemtuzumab, etc.) within 3 months of study entry

  * Patients treated with monoclonal antibodies within 3 months allowed provided disease progressed on this therapy AND no treatment received 7 days prior to study entry
  * Seven days since prior rituximab (for patients enrolled in phase I portion)
* No major surgery within 4 weeks of study entry
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-12-13 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Portlock, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- [Result] Gerecitano J, Portlock C, Hamlin P, Moskowitz CH, Noy A, Straus D, Schulman P, Dumitrescu O, Sarasohn D, Pappanicholaou J, Iasonos A, Zhang Z, Mo Q, Horanlli E, Rojas CN, Zelenetz AD, O'Connor OA. Phase I trial of weekly and twice-weekly bortezomib with rituximab, cyclophosphamide, and prednisone in relapsed or refractory non-Hodgkin lymphoma. Clin Cancer Res. 2011 Apr 15;17(8):2493-501. doi: 10.1158/1078-0432.CCR-10-1498. Epub 2011 Feb 23. PMID 21346146
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide: Phase I Weekly 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide
- 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide: Phase I Weekly 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide
- 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide: Phase I Weekly 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide
- 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide: Phase I Weekly 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide
- Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid: Phase I Twice Weekly 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide
- Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid: Phase I Twice Weekly 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide
- Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham: Phase I Twice Weekly 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide
- Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami: Phase I Twice Weekly 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide
- Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami: Phase I Twice Weekly 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide; Pegylated G-CSF
- Weekly Bortezomib Dosing Schedule: Phase II Randomized Weekly bortezomib dosing schedule
- Twice-weekly Bortezomib Dosing Schedule: Phase II Randomized Twice-weekly bortezomib dosing schedule
Period: Overall Study
Arm/Group | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Weekly Bortezomib Dosing Schedule | Twice-weekly Bortezomib Dosing Schedule
Started | 4 | 6 | 3 | 4 | 2 | 18 | 3 | 4 | 10 | 12 | 13
Completed | 4 | 6 | 3 | 4 | 2 | 18 | 3 | 4 | 10 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Weekly Bortezomib Dosing Schedule | Twice-weekly Bortezomib Dosing Schedule | Total
Number analyzed (Participants) | 4 | 6 | 3 | 4 | 2 | 18 | 3 | 4 | 10 | 12 | 13 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 1 | 2 | 0 | 10 | 1 | 3 | 9 | 6 | 6 | 42
  >=65 years | 1 | 5 | 2 | 2 | 2 | 8 | 2 | 1 | 1 | 6 | 7 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 2 | 1 | 12 | 1 | 1 | 4 | 4 | 5 | 39
  Male | 1 | 2 | 1 | 2 | 1 | 6 | 2 | 3 | 6 | 8 | 8 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  White | 4 | 6 | 3 | 3 | 0 | 17 | 2 | 3 | 8 | 11 | 11 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Maximum tolerated dose of Bortezomib in combination with Rituximab, Cyclophosphamide and Prednisone in Phase I participants
Time Frame: 2 years
Population: This outcome is only applicable for Phase I portion of the study. The purpose of the Phase I portion of the study is to determine the Maximum Tolerated Dose and for this reason the results are not separated by dose level.
Measure: Number; unit: mg/m^2 of Bortezomib
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 54 | 0
mg/m^2 of Bortezomib
  Weekly Bortezomib | 1.8 |
  Twice-Weekly Bortezomib | 1.5 |

2. Secondary Outcome: Progression-free Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of Response (Mean and Median)
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Event-free Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Toxicity of Participants Receiving Bortezomib, Rituximab, Cyclophosphamide, and Prednisone for Treatment of Non-Hodgkin's Lymphoma
Description: Toxicity assessed using NCI-CTC v. 3.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham: Phase I Twice Weekly 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide; Pegylated G-CSF
Arm/Group | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Weekly Bortezomib Dosing Schedule | Twice-weekly Bortezomib Dosing Schedule
Number analyzed (Participants) | 4 | 6 | 3 | 4 | 2 | 18 | 3 | 4 | 10 | 12 | 13
Participants | 4 | 6 | 3 | 4 | 2 | 18 | 3 | 4 | 10 | 12 | 13

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham | Weekly Bortezomib Dosing Schedule | Twice-weekly Bortezomib Dosing Schedule
All-Cause Mortality (participants affected / at risk) | 3/4 | 6/6 | 2/3 | 3/4 | 1/2 | 13/18 | 2/3 | 3/4 | 7/10 | 4/12 | 5/13
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/6 | 2/3 | 2/4 | 0/2 | 5/18 | 1/3 | 2/4 | 1/10 | 4/12 | 8/13
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 3/3 | 4/4 | 2/2 | 18/18 | 3/3 | 4/4 | 10/10 | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide (N=4) | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide (N=6) | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide (N=3) | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide (N=4) | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid (N=2) | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid (N=18) | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham (N=3) | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami (N=4) | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham (N=10) | Weekly Bortezomib Dosing Schedule (N=12) | Twice-weekly Bortezomib Dosing Schedule (N=13)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hemorrhage/Bleeding, other (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemorrhage/Bleeding assoc w/surg, intra/ post-op (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection, other (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy: sensory (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelets (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide (N=4) | 1.6 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamide (N=6) | 1.6 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide (N=3) | 1.8 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphamide (N=4) | Dose Level 1- 1.0 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid (N=2) | Dose Level 2 - 1.3 mg/m2 Bortezomib; 750 mg/m2 Cyclophosphamid (N=18) | Dose Level 3 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham (N=3) | Dose Level 4 - 1.5 mg/m2 Bortezomib; 1000 mg/m2 Cyclophosphami (N=4) | Dose Level 5 - 1.3 mg/m2 Bortezomib; 1000 mg/m2 Cyclophospham (N=10) | Weekly Bortezomib Dosing Schedule (N=12) | Twice-weekly Bortezomib Dosing Schedule (N=13)
Constipation (Gastrointestinal disorders) | 2 | 3 | 0 | 2 | 1 | 12 | 1 | 1 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 2
Fatigue (General disorders) | 2 | 3 | 2 | 2 | 0 | 10 | 1 | 1 | 4 | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4 | 0 | 6 | 1 | 3 | 3 | 5 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 2 | 0 | 3 | 0 | 0 | 2 | 3 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 2 | 0 | 5 | 0 | 1 | 3 | 6 | 2
Lymphocyte count decreased (Investigations) | 3 | 4 | 2 | 3 | 2 | 15 | 3 | 4 | 9 | 10 | 10
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 3 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 10 | 1 | 2 | 3 | 0 | 1
Platelet count decreased (Investigations) | 0 | 3 | 0 | 4 | 2 | 8 | 2 | 2 | 4 | 5 | 10
Anemia (Blood and lymphatic system disorders) | 1 | 5 | 2 | 4 | 0 | 8 | 2 | 2 | 5 | 8 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 5 | 2 | 4 | 2 | 9 | 1 | 0 | 5 | 9 | 9
White blood cell decreased (Investigations) | 2 | 4 | 2 | 4 | 2 | 9 | 1 | 2 | 5 | 10 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Fever (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INR Increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Analysis available and entered in the results section for Phase I participants. Cannot submit results on Phase II because analysis was incomplete when PI left MSK.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT00295932/Prot_SAP_000.pdf